CLINICAL TRIAL: NCT01724515
Title: PGC-1 and Mitochondrial Dysfunction in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lawrence Mandarino, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-006065 Aim 5; R01DK066483 (NIH)
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes; Obese
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Obese Non-Diabetic Subjects (Experimental): All subjects on this arm will undergo lipid infusion and muscle biopsies.
  Interventions: Other: Lipid infusion and muscle biopsies
- Type 2 Diabetic Subjects (Experimental): All subjects on this arm will undergo lipid infusion and muscle biopsies.
  Interventions: Other: Lipid infusion and muscle biopsies
- Healthy Control Subjects (Experimental): All subjects on this arm will undergo lipid infusion and muscle biopsies.
  Interventions: Other: Lipid infusion and muscle biopsies

INTERVENTIONS:
Other: Lipid infusion and muscle biopsies — Subjects will undergo a baseline muscle biopsy, a lipid infusion for 5 hours (60 ml/hr), and a muscle biopsy after the lipid infusion.

SUMMARY:
The purpose of this study is determine if you have too much fat in your body that it will decrease the conversion of food energy into energy that your body can use.

DETAILED DESCRIPTION:
The investigators' prior research has focused on defining the changes in expression of nuclear encoded mitochondrial genes that predict changes in insulin sensitivity in skeletal muscle, with the goal of defining the molecular mechanisms underlying the connection between mitochondrial dysfunction and insulin resistance in skeletal muscle.

The purpose of this study is to determine whether experimental lipid oversupply decreases mitochondrial respiratory function. We will use mitochondrial respiration studies in vitro and mass spectrometry and proteomics analysis to test the hypothesis that experimental lipid oversupply:

1. Decreases mitochondrial respiration in response to lipid fuels.
2. Reduces abundance of mitochondrial proteins.
3. Alters phosphorylation of proteins in the electron transport chain.

Three groups of subjects will be studied: lean, healthy control subjects (n=12), obese non-diabetic subjects (n=12) and patients with type 2 Diabetes Mellitus (n=12) for a total of 36 subjects. Twenty subjects have completed the study at Arizona State University; the remaining 16 subjects will be accrued at the Mayo Clinic in Arizona.

Subjects will come to the Mayo Clinic 2 times. On study Day 1 subjects will be screened with a medical history and physical exam, and a 75 g oral glucose tolerance test, measure body fat percentage, and an electrocardiogram (EKG). On Study Day 2, subjects will report to the clinic after an overnight fast. Female subjects will take a urine pregnancy test. A muscle biopsy will be performed to take a small sample from one thigh. A lipid infusion will be performed for 5 hours (60 ml/hr), with blood samples taken at 8 intervals during the infusion. At the end of the 5 hour period, a second muscle biopsy will be taken from the other thigh. The fat infusion will stop, subjects will be given lunch and allowed to leave the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Subjects may be of either sex with age as described in each protocol. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period.
3. Subjects must range in age as described in each specific protocol.
4. Subjects must have the following laboratory values:

   1. Hematocrit ≥ 35 vol%
   2. Serum creatinine ≤ 1.6 mg/dl
   3. Aspartate Aminotransferase (AST) (SGOT) < 2 times upper limit of normal
   4. Alanine Aminotransferase (ALT) (SGPT) < 2 times upper limit of normal
   5. Alkaline phosphatase < 2 times upper limit of normal
   6. Triglycerides < 150 mg/dl.
   7. Prothrombin Time (PT) 11.7 - 14.3 seconds (during Intralipid/heparin infusion, PT will be determined to insure that it is < 1.5-2.0 times the normal value.)
   8. Partial Thromboplastin Time (PTT) 23.0-37.0 seconds.

Exclusion Criteria:

1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
2. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
3. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>180, diastolic BP>105, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mitochondrial Respiration | Study Day 2, muscle biopsy approximately 6 hours after lipid infusion initiation
  Mitochondrial respiration will be measured by micropolarography.

SECONDARY OUTCOMES:
Protein Concentration of Mitochondria | Study Day 2, muscle biopsy approximately 6 hours after lipid infusion initiation
  Protein concentration will be determined by the method of Lowry. 75 micrograms of muscle lysate proteins will be separated on a 10% Sodium Dodecyl Sulfate Polyacrylamide Gel, and then visualized with Coomassie stain. The gel lane will be cut into cubes, digested with trypsin and cleaned, then protein abundance will be determined using spectral counting.
Phosphorylation of proteins | Study Day 2, muscle biopsy approximately 6 hours after lipid infusion initiation
  Phosphopeptides will be measured by mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mandarino, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States